CLINICAL TRIAL: NCT00434291
Title: A Randomized, Double-Blind, Comparative, Multi-Center Study of the Safety and Efficacy of TG-873870(Nemonoxacin) Versus Levofloxacin in Adult Patients With Community-Acquired Pneumonia (CAP)
Brief Title: Safety and Efficacy Comparison of TG-873870(Nemonoxacin) to Levofloxacin in Community-Acquired Pneumonia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TaiGen Biotechnology Co., Ltd. (Industry)
Collaborators: Quintiles, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TG-873870-02
Record Dates: First submitted 2007-02-12; First posted 2007-02-13 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Community-Acquired Pneumonia
Keywords: Community-acquired Pneumonia; fluoroquinolone; TG-873870; Nemonoxacin
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — nemonoxacin

INTERVENTIONS:
Drug: TG-873870(Nemonoxacin)

SUMMARY:
This study will test the safety and efficacy of TG-873870(Nemonoxacin) compared with Levofloxacin in adult patients with Community-Aquired Pneumonia(CAP)

DETAILED DESCRIPTION:
Community-acquired Pneumonia(CAP) remains a leading cause of death in both developing and developed countries. In the choice of antibacterial agents used to treat CAP, fluoroquinolones have received considerable attention because of their wide spectrum of bactericidal activity. TG-873870(Nemonoxacin), a non-fluorinated quinolone (NFQ), is a selective bacterial topoisomerase inhibitor. This study will test the safety and efficacy of TG-873870(Nemonoxacin) compared with Levofloxacin in adult patients with Community-Aquired Pneumonia (CAP) .

ELIGIBILITY:
Inclusion Criteria:

* If female, non-lactating and at no risk or pregnancy (post-menopausal or must use adequate birth control)
* Must be a suitable candidate for oral antibiotic therapy and must be able to swallow capsules intact
* Must have a clinical diagnosis of CAP based on clinical evidence
* Must have a chest radiograph demonstrating new or persistent/progressive infiltrates
* Must be able to produce sputum

Exclusion Criteria:

* Clinically significant conduction or other abnormality on 12-lead ECG, or QTc interval
* Patients with CAP that, in the investigator's judgment, is severe enough to require hospitalization for intravenous antibiotic therapy and/or supplemental oxygen therapy with ICU support
* Known or suspected severe bronchiectasis, cystic fibrosis, active pulmonary tuberculosis or infection with other mycobacteria or fungi, known bronchial obstruction, a history of post-obstructive pneumonia, other confounding respiratory diseases, such as lung cancer, malignancy metastatic to the lungs, lung abscess, empyema, suspected aspiration pneumonia due to vomiting, or non-bacterial respiratory infection (chronic obstructive pulmonary disease [COPD] is not exclusionary)
* Infection acquired in a hospital, nursing home, or other long-term care facility, or hospitalization for any reason within the previous 14 days
* Treatment with any antibiotics within the past 7 days prior to randomization, unless documents to be a treatment failure(72 hours treatment and not responding)
* Anticipation of the requirement for additional treatment with non-study antibacterials for any reason during the patient's participation in the study
* Treatment with chemotherapeutic agents or oncolytics during the 6 months prior to randomization or anticipated requirement for such agents during the course of the study
* Known or suspected CNS disorder that may predispose the patient to seizures or lower the seizure threshold

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2006-12; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Safety evaluation
Clinical Cure Rate

SECONDARY OUTCOMES:
Bacteriologic Cure Rate

CONTACTS AND LOCATIONS:
Overall Officials: Reury-Perng Perng, Doctor, Principal Investigator — Taipei Veterans General Hospital, Taipei, Taiwan; Ming-Lin Ho, Doctor, Principal Investigator — Chang-Hua Christian Hospital, Changhua, Taiwan; Wann-Cherng Perng, Doctor, Principal Investigator — Tri-Service General Hospital, Taipei, Taiwan; Kai-Ming Chang, Doctor, Principal Investigator — Taichung Veterans General Hospital, Taichung, Taiwan; Yen-Hsu Chen, Doctor, Principal Investigator — Kaoshiung Medical University Hospital, Kaoshiung, Taiwan; Ren-Guang Wu, Doctor, Principal Investigator — Cheng Ching Hospital, Taichung, Taiwan; Yin-Ching Chuang, Doctor, Principal Investigator — Chi-Mei Foundation Hospital, Tainan, Taiwan; Horng-Chyuan Lin, Doctor, Principal Investigator — Chang-Gung Memorial Hospital, Taoyuan, Taiwan; Yao-Kuang Wu, Doctor, Principal Investigator — Buddhist Taipei Tzu Chi General Hospital, Taipei, Taiwan; Hsi-Hsun Lin, Doctor, Principal Investigator — E-Da Hospital, Kaohsiung, Taiwan; AJ Bester, Doctor, Principal Investigator — GCT at Jubilee Hospital, RSA; J Breedt, Doctor, Principal Investigator — Bougainville Hospital, RSA; CT de Villiers, Doctor, Principal Investigator — de Villers Clinical Trials, RSA; M Gani, Doctor, Principal Investigator — GCT Trial Centre, Mercantile Hospital, RSA; Y Kelfkens, Doctor, Principal Investigator — Private, RSA; DJ Jansen van Rensburg, Doctor, Principal Investigator — Park Medical Centre, RSA; J Jurgens, Doctor, Principal Investigator — DJW Research, RSA; IH Mitha, Doctor, Principal Investigator — Benmed/Pentagon Hospital, RSA; JH Mynhardt, Doctor, Principal Investigator — Private, RSA; G Nieuwoudt, Doctor, Principal Investigator — MediTrials, RSA; J Kasumba, Doctor, Principal Investigator — JOSHA Research, RSA; E van Nieuwenhuizen, Doctor, Principal Investigator — Eastmed Clinical Trial Center, RSA; CJJ van Rensburg, Doctor, Principal Investigator — Private, RSA
Locations (20):
- South Africa (10):
  - GCT at Jubilee Hospital, Temba, North West
  - Benmed/Pentagon Hospital, Benomi
  - MediTrials, Cape Town
  - Private, Kimberley
  - DJW Research, Krugersdorp
  - GCT Trial Centre, Mercantile Hospital, Port Elizabeth
  - Private, Potchefstroom
  - Bougainville Hospital, Pretoria
  - de Villers Clinical Trials, Scottburgh
  - Park Medical Centre, Witbank
- Taiwan (10):
  - Chang-Hua Christian Hospital, Changhua
  - E-Da Hospital, Kaohsiung City
  - Kaoshiung Medical University Hospital, Kaoshiung
  - Cheng Ching Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Chi-Mei Foundation Hospital, Tainan
  - Buddhist Taipei Tzu Chi General Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang-Gung Memorial Hospital, Taoyuan District

REFERENCES:
- [Background] Bartlett JG, Breiman RF, Mandell LA, File TM Jr. Community-acquired pneumonia in adults: guidelines for management. The Infectious Diseases Society of America. Clin Infect Dis. 1998 Apr;26(4):811-38. doi: 10.1086/513953. PMID 9564457
- [Background] Mandell LA, Bartlett JG, Dowell SF, File TM Jr, Musher DM, Whitney C; Infectious Diseases Society of America. Update of practice guidelines for the management of community-acquired pneumonia in immunocompetent adults. Clin Infect Dis. 2003 Dec 1;37(11):1405-33. doi: 10.1086/380488. Epub 2003 Nov 3. No abstract available. PMID 14614663
- [Background] Bartlett JG, Dowell SF, Mandell LA, File TM Jr, Musher DM, Fine MJ. Practice guidelines for the management of community-acquired pneumonia in adults. Infectious Diseases Society of America. Clin Infect Dis. 2000 Aug;31(2):347-82. doi: 10.1086/313954. Epub 2000 Sep 7. No abstract available. PMID 10987697
- [Background] Fujimoto T, Mitsuhashi S. In vitro antibacterial activity of DR-3355, the S-(-)-isomer of ofloxacin. Chemotherapy. 1990;36(4):268-76. doi: 10.1159/000238777. PMID 2174762
- [Background] Croom KF, Goa KL. Levofloxacin: a review of its use in the treatment of bacterial infections in the United States. Drugs. 2003;63(24):2769-802. doi: 10.2165/00003495-200363240-00008. PMID 14664657
- [Background] Ellner PD, Neu HC. The inhibitory quotient. A method for interpreting minimum inhibitory concentration data. JAMA. 1981 Oct 2;246(14):1575-8. doi: 10.1001/jama.246.14.1575. PMID 7277631
- See also: NCBI — http://www.ncbi.nlm.nih.gov/